CLINICAL TRIAL: NCT05461469
Title: Safety and Feasibility of the Cornea DomeLens Ocular Surface Imaging System
Brief Title: CDL Validation Study
Status: Completed | Type: Observational
Sponsor: Occyo GmbH (Industry)
Collaborators: University Clinic for Ophthalmology and Optometry- Salzburg (Unknown)
Responsible Party: Sponsor
Other Study IDs: 2021-01-CDL
Record Dates: First submitted 2022-06-24; First posted 2022-07-18 (Actual); Last update posted 2024-04-04 (Actual); Status verified 2024-04

CONDITIONS: Eyes Dry Chronic; Chronic Conjunctivitis of Both Eyes; Limbal Stem-cell Deficiency; Eye Lesion; Eye Disease; Cataract; Eyes Dry Feeling of; Cornea Disease; Cornea Inflamed; Cornea; Injury, Abrasion; Cornea Infection
Keywords: Ocular surface; Imaging; Cornea; Conjunctiva; Dry eye disease
MeSH Terms: conditions — Limbal Stem Cell Deficiency; Cataract; Corneal Diseases; Keratitis; Corneal Injuries; Dry Eye Syndromes

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Ocular surface photography is significantly limited in standardization and reproducibility. This reduces its applicability for clinical monitoring of acute or chronic disease. The innovative lens and illumination design of the CDL system aims to yield standardized high resolution photographs of the cornea and conjunctiva as required for clinical documentation, posing a significant clinical benefit of health care providers in the field of ophthalmology.

Primary objectives: The primary objective of this study is to test the safety and feasibility of the CDL imaging system in a clinical routine setting. This will include the comparison of subjective contrast sensitivity testing post imaging, and the measurement of examination duration per imaging session, and the comparison of image lightness in mesopic versus photopic imaging.

Secondary objectives: The secondary objective of this study is to compare the image quality of the device and repeatability of lateral resolution, dynamic range, hue, saturation, lightness, and image position between colour photographs from a state-of the art slit lamp camera and the CDL system.

This is a monocentric, prospective, observational study. Patients with ocular surface disease of variable aetiology routinely assigned to ocular surface photography, following informed consent, will be imaged using state-of-the-art colour photography and the CDL imaging system. Pictures of each patient will be taken under several standardized conditions with both methods, subsequently analysed and compared by a Medical Image Processing Specialist.

DETAILED DESCRIPTION:
Number of Patients: 100 participants will be enrolled. It is expected that 80% of enrolled patients will be assessed more than once during the study period. Based on an historic analysis of ambulatory visits it is estimated that the mean overall number of study visits will be 2.6 per patient with a range from 1 to 12, resulting in an overall number of study visits of 260(100 first visits and 160 follow-up visits).

Sample size justification: The present study was designed to detect a difference in mean loss of contrast sensitivity post CDL imaging of 1 letter (letter maximum: 48) compared to slit lamp photography (mean group slit lamp 1 letter with SD 1.75, mean group CDL 2, alpha 0.05, beta 0.2, power 0.8). The resulting sample size was 96.Regarding the principal secondary endpoint of repeatability, photography will be repeated 3 times with both devices. This study design allows the conclusion on repeatability of both devices. Based on clinical experience, the investigators expect a difference in repeatability of images between the two devices of approximately 15%. With this difference the required sample size to detect a significant difference without type I or II error is 150. Incidence of not repeatable images with CDL -group 1(5%). Incidence of not repeatable images with camera slit lamp -group 2 (20%). Alpha (0.05), Beta (0.2), Power (0.8).

General Study Procedure and Assessment Schedule A clinical examination using slit lamp biomicroscopy will be undertaken by experienced cornea and ocular surface specialists. Best corrected visual acuity and contrast sensitivity will be tested. Detailed notes of the live assessment will be made of all patients using the provided case report form (CRF).This will include patient demographics (age, sex), previous ocular history, previous medical history, concomitant medication, best corrected visual acuity, history of allergies. Particular note will be made of any conjunctival, limbal or corneal abnormalities, biomicroscopic grading of conjunctival redness using Efron's grading scale, and biomicroscopic grading of corneal punctate staining using the Oxford grading scale. Imaging will be performed with a total of 12images per eye performed by one trained operator at each study visit. Of these 12 images, 6 will be taken with state of the art slit lamp photography, and 6 will be taken with the CDL system. Of the 6 images per system, three will be taken at mesopic room conditions and three at photopic room light conditions. Every series of three photographs will be timed. Any study patient who is routinely scheduled for repeated ocular surface photographs during the study period will also receive repeated CDL and slit lamp imaging at consecutive clinical visits. Following the imaging session, contrast sensitivity will be tested 30 min after the photo session. Obtained colour photographs will be anonymized, coded, and exported to a password-locked hard drive in raw format and assigned to image analysis. Any image analysis will be performed by the data and image analysis team at Occyo.

Documentation The accomplishments of the study in agreement with the EN ISO 14155-2020 guidelines, the MD and the clinical investigational plan as well as the trueness of all data documented in the CRF are the responsibility of the Investigator. All collected data of this study have to be recorded in the CRF by appropriate authorized persons. This is also valid for data of patients, who dropped-out of the study. The Investigator records the participation in a special identification list of patients. This list gives the possibility of a later identification of the patients and contains the patient number, full name, date of birth and the date of the enrolment in the study. The identification list of patients remains in the study center after the closure of the study. Additionally, the participation of the patient in this clinical study has to be recorded in the patient chart (investigational device, number of patient, start and end of the study).Further it has to be assured, that this person, who is responsible for the documentation in the CRF, can be identified. A delegation of responsibilities log with signatures and identification code of the persons, who are allowed to make entries in the CRF, will be archived in the Study Master File.

Data Recording (CRF/eCRF): First point of data entry for all study relevant parameters will be the patient file (Source data). In accordance with the clinical routine and routine data capturing, specific study related data points will be treated as direct entries in the CRF and subsequently archived according to local regulations.

Trial Folders: The trial folders should contain the complete documentation of the trial. Individually or together, they should allow the evaluation of the trial conduct and its data quality.

Trial Master File (TMF): The paper-based TMF, established at the beginning of the trial and secured in a safe place, contains all essential documents that demonstrate that the trial is conducted in accordance with regulatory requirements and ISO 14155-2020. All documents will be maintained and updated as appropriate throughout the trial. The TMF is archived at the end of the study for 15 years.

Investigator Site File (ISF): The paper-based ISF, established at the beginning of the trial will be secured in a safe place. It contains all essential documents and will be maintained by the PI(s)and delegated members of the study team. All documents will be updated as appropriate throughout the trial. Within the Monitoring, the ISF will be checked up on actuality and completeness in accordance with the formalities. After completion or discontinuation of the study this ISF has to be kept for 15 years.

Data storage Records and documents related to the study will be kept for at least 15 years Data Management The evaluation of the data takes place by the programmed range-, validity-and consistency checks. Following verification regarding the plausibility and completeness by the Monitor, data are transferred to the Sponsor, where manual/visual evaluation of the plausibility in accordance with the requirements of the EN ISO 14155-2020 is performed by the data and safety monitoring committee (quality@occyo.com).Queries may occur, which will be forwarded to the respective investigator. On the basis of the queries the Investigator has to evaluate and respond to the outlined discrepancies. For completion of the study, after the record of all entries and clarification of all queries, the database will be closed.

Statistics There will be two subgroups for statistical analysis: a) First visits b) Follow-up visits The imaging protocol will not be different for these two groups, but data from first visits will be analysed for the primary outcome parameter (safety and feasibility), while data from follow-up visits will be analysed for the secondary outcome parameters (lateral resolution, repeatability of peripheral lateral resolution, dynamic range, colour hue, saturation and lightness in different room light conditions). The difference in lightness between mesopic and photopic images will be calculated.

Procedures that take into account all the data a) Anonymization b) Digitization of paper records c) Data transfer in hard-drive to image analyst d) Analysis for completeness For the primary outcome parameter, analysis will be made as follows: The principal outcome parameter for device safety is the inter-device difference of mean intraindividual loss of contrast sensitivity. The principal outcome parameter for feasibility is the inter-device difference of examination duration for series-of-3 photographs. The outcome parameter will be tested for normal distribution and if the normality is not satisfied, normality transformations, such as log or sort, will be used. A Student t-test will be used if the data follows a normal distribution and a Wilcoxon signed rank test for nonparametric distribution. The associations between outcomes will be tested using general linear models. A level of probability of less than 0.05 will be considered statistically significant. Mean values with standard deviation will be given for normally distributed data, and medians when the normality is not satisfied. The primary outcome parameter will be correlated for analysis of repeatability using ANOVA testing.

For analysis of secondary outcome parameters, Bland-Altman analysis will be performed to assess repeatability. Examination duration for a series of 3 photographs will be timed during the imaging session and recorded.

Quality Management Training Monitoring and audits are performed for quality assurance within this clinical study. Monitoring and auditing procedures developed or endorsed by the Sponsor will be conducted, in order to comply with EN ISO 14155-2020 and local legal requirements to ensure acceptability of the study data.

Qualifications: each Investigator should be qualified by training and experience and should have adequate resources. Each individual involved in conducting a trial should be qualified by education, training and experience to perform his or her respective task(s).

Monitoring: monitoring visits by representatives of the Sponsor will be carried out to review study plan compliance, to compare CRFs and individual patient's medical records, to perform accounting of study material, and to ensure that the study is being conducted according to pertinent regulatory requirements. CRF entries will be verified with source documentation. The frequency and duration of monitoring visits will be determined according to clinical site accrual, site performance, adherence to the protocol, and data quality. Details will be presented in the Clinical Monitoring Plan. Further, the Monitor confirms that:

* the clinical investigational plan is fulfilled and deviations have to be discussed with the investigator, documented and reported to the sponsor
* the product is used complied to the clinical investigational plan and changes of the product, its application or with the clinical investigational plan have to be reported to the sponsor
* a signed and dated consent form exists for each test subject at the time of admission and before initiation
* inspection of the ISF
* documentation of the patient status
* CRF-data verification with the source data
* evaluation of the SAEs reports according to the regulations
* service and calibration of the devices are carried out and documented
* withdrawal of a test subject and/or non-compliance of the rules must be documented, discussed with the investigator and reported to the sponsor Audits and Inspections

Regulatory authorities, the ethics committees, and Sponsor's delegates may perform on-site inspections or audits, for which the Investigator must provide support at all times. During an audit following issues among other things will be inspected:

* performance of the clinical trial according to the investigation plan
* data validity
* quality of the clinical trial according to the EN ISO 14155-2020 guidelines After each external audit an audit-certificate by the auditor has to be sent to the Investigator. This certificate has to be kept in the ISF to evidence the audit to the regulatory authorities in the case of an inspection. The audit report is sent to the Sponsor of the study. An audit-certificate will be attached to the final report at the end of the study. Additionally, according to the Austrian Medical Device Law audits and inspections by regulatory authorities may be performed.

ELIGIBILITY:
Inclusion Criteria:

* Patients with ocular surface or anterior segment disease
* Written, signed and dated informed consent from the trial subject has been obtained

Exclusion Criteria:

* Current Participation in other interventional trials
* Patients unable to fixate a target
* Patients less than 18 years old
* Persons with any kind of dependency on the investigator or employed by the sponsor or investigator
* Persons held in an institution by legal or official order
* Patients with incapacity
* Pregnant or breastfeeding women

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients will be recruited from the corneal outpatient clinics of PMU. Participants will be given an information leaflet to read and a qualified and delegated physician will explain and discuss the study with the patients. If they are interested in participating, they will be asked to sign and return the study specific consent form. Every patient has the opportunity to withdraw from the study without compromise to their continued care. The reason for withdrawal from the study will be documented if volunteered. This will provide information to improve future study designs in this area of investigation.
Sampling Method: Non-Probability Sample
Enrollment: 104 (Actual)
Dates: Start 2022-04-22 (Actual); Primary Completion 2023-06-26 (Actual); Study Completion 2023-06-26 (Actual)

PRIMARY OUTCOMES:
Contrast sensitivity testing post imaging with either CDL or the slit lamp. | During the procedure
  Safety and feasibility of the CDL in clinical routine use, will be assessed by the contrast sensitivity test 30 minutes after imaging with either the CDL system or the the slit Lamp.
  Contrast sensitivity testing measures how well the eyes can distinguish between finer and finer light increments compared to dark.
  Pelli-Robson contrast sensitivity chart will be applied to the patient. This consists of rows of letters that become gradually less contrasted. They start a dark black and progress into a faint grey. The letters are on a white background. This test allows the doctor to determine the lightest contrast the patient can successfully see.
Severity and Risk of AE | up to 72 hours
  Eye damage due to illumination power exceeding applicable illumination limits -Patient discomfort from illumination-Blurred vision, after image, headache or dizziness after fixating the light target-Head trauma from bumping head against frame of device-Irritation of forehead, chin and hands which are in contact with the ophthalmic table and chin rest, following the use of disinfectants.
Severity and Risk of SAEs. | through the study completion, an average of one year
  Death, serious deterioration in the health of the subject, users, or other persons as defined by one or more of the following: a life-threatening illness or injury, or a permanent impairment of a body structure or a body functions including chronic diseases, or in-patient or prolonged hospitalization, or medical or surgical intervention to prevent life-threatening illness or injury, or permanent impairment to a body structure or a body function, fetal distress, fetal death, a congenital abnormality, or birth defect including physical or mental impairment.
Examination duration for series-of-3 photographs. | During the procedure
  The total exposure to the source of light should not exceed 7 minutes and 40seconds. The duration of taking 3 photographs of an eye will be measured.
Image lightness in mesopic versus photopic imaging. | During the procedure.
  The impact of the light in producing high quality photographs of the eye surface will be tested in mesopic room conditions (lights off) with the CDL and slit lamp and in photopic room conditions (lights on).

SECONDARY OUTCOMES:
Lateral resolution on corneal apex, limbus, and peripheral conjunctiva. | During the procedure
  Photographic lateral resolution at 2 separate locations of the limbus and peripheral conjunctiva 5mm from limbus at two clock hours in CDL vs. Slit lamp camera. The lateral resolution will be calculated from the number of pixels per capillary reference vessel of known dimension. The lateral resolution will be compared between slit lamp colour photography and the CDL imaging system. The image analysis will be done by a program developed in-house with python.
Repeatability of lateral resolution, dynamic range, hue, saturation, lightness and image position. | During the procedure
  The RGB (red, green, blue) image of the first group will be registered to the images of the second group, using affine image registration. Image registration is done to make the comparison of two images more spatially accurate. The registered RGB images will then be converted to HSL (hue, saturation, lightness) colour space and representative pixels of each image will be assessed for dynamic range, hue, saturation and lightness. The assessment will be both region based, and whole image histogram based. The image analysis will be done by a program developed in-house with python

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Ophthalmology and Optometry, Paracelsus Medical University Salzburg, Salzburg, Austria

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Ang M, Cai Y, MacPhee B, Sim DA, Keane PA, Sng CC, Egan CA, Tufail A, Larkin DF, Wilkins MR. Optical coherence tomography angiography and indocyanine green angiography for corneal vascularisation. Br J Ophthalmol. 2016 Nov;100(11):1557-1563. doi: 10.1136/bjophthalmol-2015-307706. Epub 2016 Jan 28. PMID 26823396
- [Background] Steger B, Romano V, Kaye SB. Corneal Indocyanine Green Angiography to Guide Medical and Surgical Management of Corneal Neovascularization. Cornea. 2016 Jan;35(1):41-5. doi: 10.1097/ICO.0000000000000683. PMID 26555579
- [Background] McMonnies CW, Chapman-Davies A. Assessment of conjunctival hyperemia in contact lens wearers. Part I. Am J Optom Physiol Opt. 1987 Apr;64(4):246-50. doi: 10.1097/00006324-198704000-00003. PMID 3591894
- [Background] Bron AJ, Evans VE, Smith JA. Grading of corneal and conjunctival staining in the context of other dry eye tests. Cornea. 2003 Oct;22(7):640-50. doi: 10.1097/00003226-200310000-00008. PMID 14508260
- [Background] Guthoff RF, Baudouin C, Stave J. Atlas of Confocal Laser Scanning In-Vivo Microscopy in Ophthalmology. Springer; 2007
- [Background] Krachmer JH, Mannis MJ, Holland EJ. Cornea. In: Vol I. 3rd Edition. Mosby Elsevier; 2011.
- [Background] Steger B, Romano V, Jesacher A, et al. Ocular Surface Photography 2.0 -Curved Object Plane For Corneal Imaging. Appl Opt. in press 2017
- [Background] Efron N. Grading scales for contact lens complications. Ophthalmic Physiol Opt. 1998 Mar;18(2):182-6. doi: 10.1016/s0275-5408(97)00066-5. PMID 9692040